CLINICAL TRIAL: NCT05432570
Title: Which is More Comfortable in Parotidectomy With Neuromonitoring: Using a Muscle Relaxants and Getting It Back? Not to Use it at All? Single-Blind, Prospective, Randomized Study
Brief Title: Use of Muscle Relaxants in Parotidectomy Operation With Neuromonitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, İsmail SÜMER, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Ismail03
Record Dates: First submitted 2022-06-19; First posted 2022-06-27 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Intubation; Difficult or Failed; Muscle Relaxation; Anesthesia Intubation Complication; Airway Complication of Anesthesia
Keywords: parotid surgery; muscle relaxants; airway management; neuromonitoring
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Before the operation, the appropriate anesthesia approach will be selected for the randomized patient group and anesthesia management will be performed according to the selected group. The surgeon who will perform the operation will perform the operation without knowing which method is chosen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Muscle Relaxants Used (Active Comparator): Muscle Relaxants Used
  Interventions: Procedure: Group A - Muscle Relaxants Used
- Group B - No Muscle Relaxants (Active Comparator): No Muscle Relaxants
  Interventions: Procedure: Group B - No Muscle Relaxants

INTERVENTIONS:
Procedure: Group A - Muscle Relaxants Used — Induction will be achieved with 1 mg/kg lidocaine, 2 μg/kg fentanyl, 2 mg/kg propofol, and 0.6 mg/kg rocuronium stored at 4 degrees. After the induction, laryngoscopy will be performed with a Macintosh laryngoscope after 2 minutes of manual ventilation after muscle relaxant by an anesthesiologist with at least 4 years of experience. It will be intubated with a tube with an inner diameter of 8 mm for men and 7 mm for women. The cuff of the intubation tube will be connected to a manometer and inflated at a pressure of 20-30 mmHg until there is no air leak. Intubation will be confirmed by the appearance of end-tidal CO2.
  Arms: Group A - Muscle Relaxants Used
Procedure: Group B - No Muscle Relaxants — Induction will be provided with 1 mg/kg lidocaine, 2 μg/kg fentanyl, 2 mg/kg propofol. After ventilation, vocal cords will be seen with a Macintosh laryngoscope, and 2cc of 2% lidocaine will be applied to the vocal cords as a spray with the help of a 5 ml injector. After ventilation, laryngoscopy will be performed with a Macintosh laryngoscope by an anesthesiologist with at least 4 years of experience. It will be intubated with a tube with an inner diameter of 8 mm for men and 7 mm for women. The cuff of the intubation tube will be connected to a manometer and inflated at a pressure of 20-30 mmHg until there is no air leak. Intubation will be confirmed by the appearance of end-tidal CO2.
  Arms: Group B - No Muscle Relaxants

SUMMARY:
Neuromuscular blockers provide muscle relaxation by blocking the electrical conduction to motor nerves and facilitate endotracheal tube placement while relaxing the whole body for surgical comfort during general anesthesia. Parotid surgery is a procedure performed by ear, nose and throat physicians, and as a complication during this procedure, permanent facial paralysis may develop due to damage to the facial nerve. Intraoperative nerve monitoring is frequently used to avoid this complication. The application of local anesthetic to the vocal cords and into the trachea has been tried and found useful for induction of anesthesia without the use of neuromuscular blockers. In studies conducted with this technique, a standard local anesthetic dose was not specified and local anesthetics were generally administered alone and in high doses. It is expected that anesthesia induction and intubation without the use of muscle relaxants will not affect the comfort of the patient and the procedure, but will increase the surgical time and surgical satisfaction.

DETAILED DESCRIPTION:
A general anesthesia technique is required, which will not only facilitate tracheal intubation during anesthesia but also minimize complications that may develop during and after surgery and/or anesthesia without the neuromuscular blocker effect. For this purpose; Induction techniques can be used without the use of muscle relaxants, which will affect the hemodynamic response less. By applying muscle relaxants, its effect can be expected to disappear completely during surgery, or muscle relaxants such as succinylcholine, which are very short-acting, can be used. However, the use of succinylcholine has almost ceased to be used clinically due to anaphylaxis, severe post-operative muscle pain, increased serum potassium levels, rarely prolonged effects, and other cardiovascular side effects that may develop. Sugammadex, which has recently entered clinical use, can be used to reverse the effect of muscle relaxants. After induction, it is necessary to use high doses of sugammadex to immediately reverse the muscle relaxant effect. Waiting for the effects of muscle relaxants to pass, especially in surgical procedures that require neuromonitoring, prolongs the surgical time. This again leads to high costs. The application of local anesthetic to the vocal cords and into the trachea has been tried and found useful for induction of anesthesia without the use of neuromuscular blockers. In studies conducted with this technique, a standard local anesthetic dose was not specified and local anesthetics were generally administered alone and in high doses. Therefore, local anesthetic administered together with the inhalation agent during induction may provide better comfort during tracheal intubation. It is expected that anesthesia induction and intubation without the use of muscle relaxants will not affect the comfort of the patient and the procedure, but will increase the surgical time and surgical satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Age between 18-65y
* Mallampati 1-2
* Patients who will undergo elective paratidectomy

Exclusion Criteria:

* History of head and neck surgery
* Body mass index less than 19 or greater than 30
* Muscle relaxant allergy
* Lidocaine allergy
* IDS score >5
* Patients whose hunger is not suitable
* Uncontrolled hypertension, bronchial asthma, tracheal pathology
* undergoing emergency surgery
* Cases that cannot give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Difficulty of Intubation | during intubation after induction of anesthesia
  The intubation difficulty scale (IDS) of patients will be used to determine the difficulty of intubation during laryngoscopy, and the Helbo-Hansen scoring system-Steyn Modification will be used to determine the quality of laryngoscopy.
  Intubation Difficulty Scale (IDS) score, which is a function of seven parameters, resulting in a progressive, quantitative determination of intubation complexity.
  intubation difficulty may be defined as a measure of the degree of divergence from a predefined "ideal" intubation, i.e., one performed without effort, on the first attempt, practiced by one operator, using one technique, with full visualization of the laryngeal aperture and vocal cords abducted. Such an intubation is accorded an IDS value of 0. Each variation from this defined "ideal" intubation increases the degree of difficulty, the overall score being the sum of all variations from this definition. Impossible intubation is defined by infinity (IDS =[infinity]).
Difficulty of Laryngoscopy | during intubation after induction of anesthesia
  The Helbo-Hansen scoring system-Steyn Modification will be used to determine the quality of laryngoscopy.
  Helbo-Hensen et al. with Steyn modification includes five criteria; ease of laryngoscopy, degree of coughing, position of vocal cords, jaw relaxation, and limb movement and graded on a 4-point scale.Total score of 5 will considere to be excellent, 6-10 good, 11-15 poor, and 16-20 bad. Total scores will divide into clinically acceptable and not acceptable scores (total score ≤ 10 acceptable, >10 unacceptable).
Number of Intubation Attempts | during intubation after induction of anesthesia]
  The number of intubation attempts between both groups will be recorded. that patients are intubated will be confirmed by the presence of end tidal carbon dioxide.

SECONDARY OUTCOMES:
Sore throat | up to 24 hours postoperative period
  Sore throat of the patients was evaluated as present or absent at the postoperative 30th minute, 2,6 and 24 hours by the patient.
Dysphagia | up to 24 hours postoperative period
  Dysphagia of the patients was evaluated as present or absent at the postoperative 30th minute, 2,6 and 24 hours by the patient.
Laryngospasm | up to 24 hours postoperative period
  Laryngospasm of the patients was evaluated as present or absent at the postoperative 30th minute, 2,6 and 24 hours by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Sumer, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)